CLINICAL TRIAL: NCT05624203
Title: Clinical Efficacy of Extracorporeal Cardiac Shock Wave Therapy in Patients With Ischemia-reperfusion Injury
Acronym: CEECSWIRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Xian-bin li, Principal Investigator, First Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1stKunmingMCYN
Record Dates: First submitted 2022-11-03; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Reperfusion Injury; Treatment Outcome; Prognosis; ST Elevation Myocardial Infarction
Keywords: extracorporeal cardiac shock waves; Endothelial progenitor cell; miR-140-3p
MeSH Terms: conditions — Myocardial Reperfusion Injury; ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Patients with acute ST-segment elevation myocardial infarction undergoing Percutaneous coronary intervention (PCI) were randomly divided into extracorporeal cardiac shock wave treatment group and blank control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extracorporeal cardiac shock wave therapy was performed（ECSW） (Experimental): Patients with acute ST-segment elevation myocardial infarction who underwent Percutaneous coronary intervention (PCI) were treated with extracorporeal cardiac shock wave therapy 2-3 days after operation. The duration of treatment was 3 months, and 9 treatments were completed within 3 months as a course. One week of treatment was followed by a 3-week rest in each month. CSWT was performed three times in each treatment week, respectively on the 1st, 3rd, and 5th day of the treatment week, for a total of 3 months.
  Interventions: Device: Extracorporeal cardiac shock wave therapy(ECSW)
- Extracorporeal cardiac shock wave therapy was not performed（NO ECSW） (No Intervention): Patients with acute ST-segment elevation myocardial infarction undergoing Percutaneous coronary intervention (PCI) are not treated with extracorporeal cardiac shock wave

INTERVENTIONS:
Device: Extracorporeal cardiac shock wave therapy(ECSW) — Extracorporeal cardiac shock wave therapy (CSWT) is a cutting-edge technology developed in the world for more than 20 years. It is mainly used in the treatment of refractory angina pectoris of coronary heart disease. The mechanism of extracorporeal cardiac shock wave therapy is mainly due to the small attenuation, small shear stress and strong penetration force of shock wave when propagating in human tissues. Shear stress and hole effect are generated in the focal area of shock wave, which leads to the repeated formation/rupture of microbubbles in tissue/cell microenvironment, resulting in various physical and biological effects. These physical mechanisms trigger a series of biological effects, such as promoting the expression of various intracellular cytokines and angiogenic factors, activating related signal transduction pathways, inhibiting apoptosis and oxidative stress, and finally increasing the number of new blood vessels in the treatment area and improving the ischemic state.
  Arms: Extracorporeal cardiac shock wave therapy was performed（ECSW）

SUMMARY:
This trial was a prospective, open-label, single-center, randomized trial, To observe the clinical efficacy of extracorporeal cardiac shock wave in the treatment of patients with myocardial ischemia-reperfusion injury and the difference in the level of endothelial progenitor cell-derived miR-140-3p in patients with myocardial ischemia-reperfusion injury treated with extracorporeal cardiac shock wave and control group and its relationship with clinical efficacy and prognosis. In order to provide a new therapy for patients with myocardial ischemia-reperfusion injury.

DETAILED DESCRIPTION:
This trial was a prospective, open-label, single-center, randomized trial, To observe the clinical efficacy of extracorporeal cardiac shock wave in the treatment of patients with myocardial ischemia-reperfusion injury and the difference in the level of endothelial progenitor cell-derived miR-140-3p in patients with myocardial ischemia-reperfusion injury treated with extracorporeal cardiac shock wave and control group and its relationship with clinical efficacy and prognosis. In order to provide a new therapy for patients with myocardial ischemia-reperfusion injury.Patients with acute ST-segment elevation myocardial infarction who underwent coronary artery stenting (PCI) were randomly divided into extracorporeal cardiac shock wave treatment group and blank control group. The primary endpoint was to analyze the clinical symptoms, cardiac structure and function, coronary microcirculation, readmission rate, related score and prognosis between the two groups. The secondary end point was to draw the survival curve of the two groups according to the follow-up situation, and establish a Cox regression model to analyze whether the survival prognosis of patients was correlated with the expression level of miR-140-3p.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years The patient was diagnosed with acute ST-segment elevation myocardial infarction for the first time, and coronary angiography showed moderate to severe coronary artery stenosis. PCI was performed within 12 hours of the onset of the disease according to the current guidelines, and postoperative hemodynamic stability was achieved CCS angina pectoris grade Ⅱ or above, NYHA cardiac function grade I-Ⅲ Imaging examination [stress echocardiography and/or stress myocardial perfusion imaging] suggested objective evidence of reversible myocardial ischemia Voluntary participation, able to cooperate with treatment and follow-up, signed informed consent.

Exclusion Criteria:

severe unprotected left main stem lesions Left ventricular systolic function was impaired with hemodynamic instability chronic obstructive pulmonary disease, pulmonary maculopathy, post-pseudobulbar placement or other causes of poor sonographic window Combined with chest malignant tumor pregnancy The skin of the treatment area is broken or infected NYHA cardiac function grade Ⅳ Acute myocarditis, pericarditis, moderate or large amount of pericardial effusion, infective endocarditis, deep vein thrombosis, intracardiac thrombosis; Severe aortic stenosis, aortic aneurysm, thoracic aortic dissection, thoracic aortic aneurysm, after heart transplantation, metal heart valve replacement, pulmonary embolism patients undergoing thrombolysis and surgical bypass Patients with a history of mental illness, poor compliance and inability to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
A composite of death, myocardial infarction, or cerebrovascular events | 24months
  24 months after the index procedure

SECONDARY OUTCOMES:
Expression level of miR-140-3p | 1, 2, 3, 6, 12 and 24 months
  The expression levels of miR-140-3p in exosomes derived from endothelial progenitor cells (EPCs) were measured in peripheral blood collected from patients at 1, 2, 3, 6, 12 and 24 months
All cause Death | 2 years
  All-cause mortality 2 years after surgery
cardiac death | 2 years
  Cardiac death 2 years after surgery
Myocardial infarction (MI) | 2 years
  Myocardial infarction 2 years after surgery
Cerebrovascular accident (CVA) | 2 years
  Cerebrovascular accident 2 years after surgery
Major adverse cardiocerebral event (MACCE): death, MI, CVA, or any revascularization | 2 years
  Major adverse cardiac and cerebral events 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cai Hongyan, Dr., Study Director — First Affiliated Hospital of Kunming Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Bulluck H, Yellon DM, Hausenloy DJ. Reducing myocardial infarct size: challenges and future opportunities. Heart. 2016 Mar;102(5):341-8. doi: 10.1136/heartjnl-2015-307855. Epub 2015 Dec 16. PMID 26674987
- [Background] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Background] Sahoo S, Klychko E, Thorne T, Misener S, Schultz KM, Millay M, Ito A, Liu T, Kamide C, Agrawal H, Perlman H, Qin G, Kishore R, Losordo DW. Exosomes from human CD34(+) stem cells mediate their proangiogenic paracrine activity. Circ Res. 2011 Sep 16;109(7):724-8. doi: 10.1161/CIRCRESAHA.111.253286. Epub 2011 Aug 11. PMID 21835908
- [Background] Arslan F, Lai RC, Smeets MB, Akeroyd L, Choo A, Aguor EN, Timmers L, van Rijen HV, Doevendans PA, Pasterkamp G, Lim SK, de Kleijn DP. Mesenchymal stem cell-derived exosomes increase ATP levels, decrease oxidative stress and activate PI3K/Akt pathway to enhance myocardial viability and prevent adverse remodeling after myocardial ischemia/reperfusion injury. Stem Cell Res. 2013 May;10(3):301-12. doi: 10.1016/j.scr.2013.01.002. Epub 2013 Jan 14. PMID 23399448
- [Background] Kooijmans SA, Vader P, van Dommelen SM, van Solinge WW, Schiffelers RM. Exosome mimetics: a novel class of drug delivery systems. Int J Nanomedicine. 2012;7:1525-41. doi: 10.2147/IJN.S29661. Epub 2012 Mar 16. PMID 22619510
- [Background] Feng Y, Huang W, Wani M, Yu X, Ashraf M. Ischemic preconditioning potentiates the protective effect of stem cells through secretion of exosomes by targeting Mecp2 via miR-22. PLoS One. 2014 Feb 18;9(2):e88685. doi: 10.1371/journal.pone.0088685. eCollection 2014. PMID 24558412
- [Background] Gollmann-Tepekoylu C, Polzl L, Graber M, Hirsch J, Nagele F, Lobenwein D, Hess MW, Blumer MJ, Kirchmair E, Zipperle J, Hromada C, Muhleder S, Hackl H, Hermann M, Al Khamisi H, Forster M, Lichtenauer M, Mittermayr R, Paulus P, Fritsch H, Bonaros N, Kirchmair R, Sluijter JPG, Davidson S, Grimm M, Holfeld J. miR-19a-3p containing exosomes improve function of ischaemic myocardium upon shock wave therapy. Cardiovasc Res. 2020 May 1;116(6):1226-1236. doi: 10.1093/cvr/cvz209. PMID 31410448
- [Background] Kikuchi Y, Ito K, Shindo T, Hao K, Shiroto T, Matsumoto Y, Takahashi J, Matsubara T, Yamada A, Ozaki Y, Hiroe M, Misumi K, Ota H, Takanami K, Hiraide T, Takase K, Tanji F, Tomata Y, Tsuji I, Shimokawa H. A multicenter trial of extracorporeal cardiac shock wave therapy for refractory angina pectoris: report of the highly advanced medical treatment in Japan. Heart Vessels. 2019 Jan;34(1):104-113. doi: 10.1007/s00380-018-1215-4. Epub 2018 Jun 25. PMID 29942978
- [Background] Kagaya Y, Ito K, Takahashi J, Matsumoto Y, Shiroto T, Tsuburaya R, Kikuchi Y, Hao K, Nishimiya K, Shindo T, Ogata T, Kurosawa R, Eguchi K, Monma Y, Ichijo S, Hatanaka K, Miyata S, Shimokawa H. Low-energy cardiac shockwave therapy to suppress left ventricular remodeling in patients with acute myocardial infarction: a first-in-human study. Coron Artery Dis. 2018 Jun;29(4):294-300. doi: 10.1097/MCA.0000000000000577. PMID 29068804
- [Background] Cai HY, Li L, Guo T, Wang YU, Ma TK, Xiao JM, Zhao L, Fang Y, Yang P, Zhao HU. Cardiac shockwave therapy improves myocardial function in patients with refractory coronary artery disease by promoting VEGF and IL-8 secretion to mediate the proliferation of endothelial progenitor cells. Exp Ther Med. 2015 Dec;10(6):2410-2416. doi: 10.3892/etm.2015.2820. Epub 2015 Oct 20. PMID 26668649
- [Background] Yang D, Wang M, Hu Z, Ma Y, Shi Y, Cao X, Guo T, Cai H, Cai H. Extracorporeal Cardiac Shock Wave-Induced Exosome Derived From Endothelial Colony-Forming Cells Carrying miR-140-3p Alleviate Cardiomyocyte Hypoxia/Reoxygenation Injury via the PTEN/PI3K/AKT Pathway. Front Cell Dev Biol. 2022 Jan 10;9:779936. doi: 10.3389/fcell.2021.779936. eCollection 2021. PMID 35083214
- [Derived] Li X, Zhang C, Liu C, Ma Y, Shi Y, Ye Y, Ma X, Liu Y, Luo X, Lin F, Wang J, Tao J, Lun J, Cai H, Hu Z. Principle and design of clinical efficacy observation of extracorporeal cardiac shock wave therapy for patients with myocardial ischemia-reperfusion injury: A prospective randomized controlled trial protocol. PLoS One. 2023 Dec 8;18(12):e0294060. doi: 10.1371/journal.pone.0294060. eCollection 2023. PMID 38064454